CLINICAL TRIAL: NCT01811888
Title: Painful Knee Prosthesis. Relationship Between Endogenous Analgesia and Persistent Post Surgical Pain.
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, CDursteler, MD, Parc de Salut Mar
Other Study IDs: TKAPAIN
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with knee osteoarthritis
  Interventions: Behavioral: Quantitative sensory testing (QST)

INTERVENTIONS:
Behavioral: Quantitative sensory testing (QST)

SUMMARY:
This is a prospective, observational study, aimed to establish the relationship between an inefficient endogenous pain modulation before surgery (total knee arthroplasty; TKA) and the probability to develop chronic pain after surgery (persistent post surgical pain). Endogenous analgesia efficiency will be measured during the month previous to surgery using quantitative sensory testing (QST). Persistent post surgical pain will be defined as presence of pain in movement greater than 3 points in a 0-10 numerical scale in the operated knee, 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 patients
* Scheduled for primary total knee arthroplasty
* Disposition to visits and scheduled tests

Exclusion Criteria:

* Previous surgery on knee to be operated
* Documented peripheral neuropathy
* Severe disease or condition that could potentially interfere with interpretation of tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis scheduled for total knee artheroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Presence of pain in the operated knee, 6 months after surgery. | Presence of pain greater than 3 points in a 0-10 numerical scale in the operated knee, 6 months after surgery.

SECONDARY OUTCOMES:
Endogenous Analgesia efficiency measured with QST (Quantitative sensory testing) techniques. | From start of recruitment untill day 180.

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio d'Anestesia i Reanimació, Hospital del Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Dursteler C, Salazar Y, Rodriguez U, Pelfort X, Verdie LP. Conditioned pain modulation predicts persistent pain after knee replacement surgery. Pain Rep. 2021 Mar 29;6(1):e910. doi: 10.1097/PR9.0000000000000910. eCollection 2021 Jan-Feb. PMID 33817538